CLINICAL TRIAL: NCT01528228
Title: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) on Postoperative Pain and Function Following Arthroscopic Knee Surgery: A Prospective Randomized Clinical Trial Pilot Study
Brief Title: Effects of TENS Therapy Following Arthroscopic Knee Surgery
Acronym: TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TENS Study #110518-001
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured TENS Therapy (Active Comparator): This group will be given an active TENS unit to use.
  Interventions: Device: TENS Treatment with functional or disabled unit
- Sham TENS Therapy (Sham Comparator): This group will receive a placebo TENS unit which has been functionally disabled to provide a short initial electrical impulse then cease delivering that impulse.
  Interventions: Device: TENS Treatment with functional or disabled unit

INTERVENTIONS:
Device: TENS Treatment with functional or disabled unit — TENS treatment will be standardized and will consist of 20 minute sessions three times per day at the manufacturer's recommended settings for both functional and disabled TENS units.
  Other Names: EMPI Select Pain Control System

SUMMARY:
Following standard of care procedures for arthroscopy knee surgery it is anticipated that Transcutaneous Electrical Nerve Stimulation (TENS) will provide improved pain relief and improve functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* BMI<50
* No significant joint malalignment
* No significant ligamentous instability
* No significant radiographic joint space narrowing
* No prior significant knee surgery
* Unilateral knee surgery
* Not workman's compensation
* Planned knee arthroscopy for meniscectomy, chondroplasty or synovectomy

Exclusion Criteria:

* Age <18 or >60
* BMI > 50
* Significant joint malalignment
* Significant ligamentous instability
* Significant radiographic joint space narrowing
* Prior significant knee surgery
* Bilateral knee surgery planned
* Worker's Compensation
* No planned knee arthroscopy for menisectomy, chondroplasty or synovectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07-01; Primary Completion 2012-04-01 (Actual); Study Completion 2012-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Marberry, MD, Principal Investigator — A.T. Still University
Locations (1):
- North Missouri Sports Medicine and Orthopaedic Surgery, Kirksville, Missouri, United States

REFERENCES:
- [Background] Breit R, Van der Wall H. Transcutaneous electrical nerve stimulation for postoperative pain relief after total knee arthroplasty. J Arthroplasty. 2004 Jan;19(1):45-8. doi: 10.1016/s0883-5403(03)00458-3. PMID 14716650
- [Background] Lewek M, Stevens J, Snyder-Mackler L. The use of electrical stimulation to increase quadriceps femoris muscle force in an elderly patient following a total knee arthroplasty. Phys Ther. 2001 Sep;81(9):1565-71. doi: 10.1093/ptj/81.9.1565. PMID 11688592
- [Background] Paternostro-Sluga T, Fialka C, Alacamliogliu Y, Saradeth T, Fialka-Moser V. Neuromuscular electrical stimulation after anterior cruciate ligament surgery. Clin Orthop Relat Res. 1999 Nov;(368):166-75. PMID 10613165
- [Background] Wang B, Tang J, White PF, Naruse R, Sloninsky A, Kariger R, Gold J, Wender RH. Effect of the intensity of transcutaneous acupoint electrical stimulation on the postoperative analgesic requirement. Anesth Analg. 1997 Aug;85(2):406-13. doi: 10.1097/00000539-199708000-00029. PMID 9249122
- [Background] Hargreaves A, Lander J. Use of transcutaneous electrical nerve stimulation for postoperative pain. Nurs Res. 1989 May-Jun;38(3):159-61. PMID 2785684
- [Background] Arvidsson I, Eriksson E. Postoperative TENS pain relief after knee surgery: objective evaluation. Orthopedics. 1986 Oct;9(10):1346-51. doi: 10.3928/0147-7447-19861001-06. PMID 3490659
- [Background] Tyler E, Caldwell C, Ghia JN. Transcutaneous electrical nerve stimulation: an alternative approach to the management of postoperative pain. Anesth Analg. 1982 May;61(5):449-56. No abstract available. PMID 6175251
- [Background] Neary JM. Transcutaneous electrical nerve stimulation for the relief of post-incisional surgical pain. AANA J. 1981 Apr;49(2):151-5. No abstract available. PMID 6111884
- [Background] Cooperman AM, Hall B, Mikalacki K, Hardy R, Sardar E. Use of transcutaneous electrical stimulation in the control of postoperative pain. Am J Surg. 1977 Feb;133(2):185-7. doi: 10.1016/0002-9610(77)90077-0. PMID 319697
- [Background] Selfe TK, Taylor AG. Acupuncture and osteoarthritis of the knee: a review of randomized, controlled trials. Fam Community Health. 2008 Jul-Sep;31(3):247-54. doi: 10.1097/01.FCH.0000324482.78577.0f. PMID 18552606
- [Background] Eyigor S, Karapolat H, Ibisoglu U, Durmaz B. [Does transcutaneous electrical nerve stimulation or therapeutic ultrasound increase the effectiveness of exercise for knee osteoarthritis: a randomized controlled study]. Agri. 2008 Jan;20(1):32-40. Turkish. PMID 18338277
- [Background] Cetin N, Aytar A, Atalay A, Akman MN. Comparing hot pack, short-wave diathermy, ultrasound, and TENS on isokinetic strength, pain, and functional status of women with osteoarthritic knees: a single-blind, randomized, controlled trial. Am J Phys Med Rehabil. 2008 Jun;87(6):443-51. doi: 10.1097/PHM.0b013e318174e467. PMID 18496246
- [Background] Burch FX, Tarro JN, Greenberg JJ, Carroll WJ. Evaluating the benefits of patterned stimulation in the treatment of osteoarthritis of the knee: a multi-center, randomized, single-blind, controlled study with an independent masked evaluator. Osteoarthritis Cartilage. 2008 Aug;16(8):865-72. doi: 10.1016/j.joca.2007.11.013. Epub 2008 Feb 8. PMID 18262443
- [Background] Kang RW, Lewis PB, Kramer A, Hayden JK, Cole BJ. Prospective randomized single-blinded controlled clinical trial of percutaneous neuromodulation pain therapy device versus sham for the osteoarthritic knee: a pilot study. Orthopedics. 2007 Jun;30(6):439-45. doi: 10.3928/01477447-20070601-11. No abstract available. PMID 17598487
- [Background] Paker N, Tekdos D, Kesiktas N, Soy D. Comparison of the therapeutic efficacy of TENS versus intra-articular hyaluronic acid injection in patients with knee osteoarthritis: a prospective randomized study. Adv Ther. 2006 Mar-Apr;23(2):342-53. doi: 10.1007/BF02850139. PMID 16751166
- [Background] Bjordal JM, Lopes-Martins RA, Bogen B, Johnson M. Physical treatments have valuable role in osteoarthritis. BMJ. 2006 Apr 8;332(7545):853. doi: 10.1136/bmj.332.7545.853. No abstract available. PMID 16601058
- [Background] Casimiro L, Barnsley L, Brosseau L, Milne S, Robinson VA, Tugwell P, Wells G. Acupuncture and electroacupuncture for the treatment of rheumatoid arthritis. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD003788. doi: 10.1002/14651858.CD003788.pub2. PMID 16235342
- [Background] Law PP, Cheing GL, Tsui AY. Does transcutaneous electrical nerve stimulation improve the physical performance of people with knee osteoarthritis? J Clin Rheumatol. 2004 Dec;10(6):295-9. doi: 10.1097/01.rhu.0000147047.77460.b0. PMID 17043536
- [Background] Law PP, Cheing GL. Optimal stimulation frequency of transcutaneous electrical nerve stimulation on people with knee osteoarthritis. J Rehabil Med. 2004 Sep;36(5):220-5. doi: 10.1080/16501970410029834. PMID 15626162
- [Background] Cheing GL, Hui-Chan CW. Would the addition of TENS to exercise training produce better physical performance outcomes in people with knee osteoarthritis than either intervention alone? Clin Rehabil. 2004 Aug;18(5):487-97. doi: 10.1191/0269215504cr760oa. PMID 15293483
- [Background] Talbot LA, Gaines JM, Ling SM, Metter EJ. A home-based protocol of electrical muscle stimulation for quadriceps muscle strength in older adults with osteoarthritis of the knee. J Rheumatol. 2003 Jul;30(7):1571-8. PMID 12858461
- [Background] Cheing GL, Tsui AY, Lo SK, Hui-Chan CW. Optimal stimulation duration of tens in the management of osteoarthritic knee pain. J Rehabil Med. 2003 Mar;35(2):62-8. doi: 10.1080/16501970306116. PMID 12691335
- [Background] Hopkins J, Ingersoll CD, Edwards J, Klootwyk TE. Cryotherapy and Transcutaneous Electric Neuromuscular Stimulation Decrease Arthrogenic Muscle Inhibition of the Vastus Medialis After Knee Joint Effusion. J Athl Train. 2002 Mar;37(1):25-31. PMID 12937440
- [Background] Cheing GL, Hui-Chan CW, Chan KM. Does four weeks of TENS and/or isometric exercise produce cumulative reduction of osteoarthritic knee pain? Clin Rehabil. 2002 Nov;16(7):749-60. doi: 10.1191/0269215502cr549oa. PMID 12428824
- [Background] Osiri M, Welch V, Brosseau L, Shea B, McGowan J, Tugwell P, Wells G. Transcutaneous electrical nerve stimulation for knee osteoarthritis. Cochrane Database Syst Rev. 2000;(4):CD002823. doi: 10.1002/14651858.CD002823. PMID 11034768
- [Background] Yurtkuran M, Kocagil T. TENS, electroacupuncture and ice massage: comparison of treatment for osteoarthritis of the knee. Am J Acupunct. 1999;27(3-4):133-40. PMID 10729968
- [Background] Brandt KD. The importance of nonpharmacologic approaches in management of osteoarthritis. Am J Med. 1998 Jul 27;105(1B):39S-44S. doi: 10.1016/s0002-9343(98)00075-8. PMID 9715833
- [Background] Hunt SA, Jazrawi LM, Sherman OH. Arthroscopic management of osteoarthritis of the knee. J Am Acad Orthop Surg. 2002 Sep-Oct;10(5):356-63. doi: 10.5435/00124635-200209000-00007. PMID 12374486
- [Background] Taylor P, Hallett M, Flaherty L. Treatment of osteoarthritis of the knee with transcutaneous electrical nerve stimulation. Pain. 1981 Oct;11(2):233-240. doi: 10.1016/0304-3959(81)90008-7. PMID 7033891
- [Background] Drosos GI, Stavropoulos NI, Katsis A, Kesidis K, Kazakos K, Verettas DA. Post-operative pain after knee arthroscopy and related factors. Open Orthop J. 2008 Jun 13;2:110-4. doi: 10.2174/1874325000802010110. PMID 19478890
- [Background] Sinatra RS, Torres J, Bustos AM. Pain management after major orthopaedic surgery: current strategies and new concepts. J Am Acad Orthop Surg. 2002 Mar-Apr;10(2):117-29. doi: 10.5435/00124635-200203000-00007. PMID 11929206
- [Background] Phillips WJ, Currier BL. Analgesic pharmacology: II. Specific analgesics. J Am Acad Orthop Surg. 2004 Jul-Aug;12(4):221-33. doi: 10.5435/00124635-200407000-00003. PMID 15473674
- [Background] Phillips WJ, Currier BL. Analgesic pharmacology: I. Neurophysiology. J Am Acad Orthop Surg. 2004 Jul-Aug;12(4):213-20. doi: 10.5435/00124635-200407000-00002. PMID 15473673
- [Background] Suzuki M, Yamada S, Inamura A, Omori Y, Kirimoto H, Sugimura S, Miyamoto M. Reliability and validity of measurements of knee extension strength obtained from nursing home residents with dementia. Am J Phys Med Rehabil. 2009 Nov;88(11):924-33. doi: 10.1097/PHM.0b013e3181ae1003. PMID 19661779
- [Background] Mahony K, Hunt A, Daley D, Sims S, Adams R. Inter-tester reliability and precision of manual muscle testing and hand-held dynamometry in lower limb muscles of children with spina bifida. Phys Occup Ther Pediatr. 2009;29(1):44-59. doi: 10.1080/01942630802574858. PMID 19197758
- [Background] Katz-Leurer M, Rottem H, Meyer S. Hand-held dynamometry in children with traumatic brain injury: within-session reliability. Pediatr Phys Ther. 2008 Fall;20(3):259-63. doi: 10.1097/PEP.0b013e3181824782. PMID 18703964
- [Background] Bell DR, Padua DA, Clark MA. Muscle strength and flexibility characteristics of people displaying excessive medial knee displacement. Arch Phys Med Rehabil. 2008 Jul;89(7):1323-8. doi: 10.1016/j.apmr.2007.11.048. PMID 18586134
- [Background] Lu TW, Hsu HC, Chang LY, Chen HL. Enhancing the examiner's resisting force improves the reliability of manual muscle strength measurements: comparison of a new device with hand-held dynamometry. J Rehabil Med. 2007 Nov;39(9):679-84. doi: 10.2340/16501977-0107. PMID 17999004
- [Background] Crompton J, Galea MP, Phillips B. Hand-held dynamometry for muscle strength measurement in children with cerebral palsy. Dev Med Child Neurol. 2007 Feb;49(2):106-11. doi: 10.1111/j.1469-8749.2007.00106.x. PMID 17253996
- [Background] O'Shea SD, Taylor NF, Paratz JD. Measuring muscle strength for people with chronic obstructive pulmonary disease: retest reliability of hand-held dynamometry. Arch Phys Med Rehabil. 2007 Jan;88(1):32-6. doi: 10.1016/j.apmr.2006.10.002. PMID 17207672
- [Background] Bohannon RW. Hand-held dynamometry: adoption 1900-2005. Percept Mot Skills. 2006 Aug;103(1):3-4. doi: 10.2466/pms.103.1.3-4. PMID 17037637
- [Background] Li RC, Jasiewicz JM, Middleton J, Condie P, Barriskill A, Hebnes H, Purcell B. The development, validity, and reliability of a manual muscle testing device with integrated limb position sensors. Arch Phys Med Rehabil. 2006 Mar;87(3):411-7. doi: 10.1016/j.apmr.2005.11.011. PMID 16500178
- [Background] Roy MA, Doherty TJ. Reliability of hand-held dynamometry in assessment of knee extensor strength after hip fracture. Am J Phys Med Rehabil. 2004 Nov;83(11):813-8. doi: 10.1097/01.phm.0000143405.17932.78. PMID 15502733
- [Background] Piao C, Yoshimoto N, Shitama H, Makino K, Wada F, Hachisuka K. Validity and reliability of the measurement of the quardriceps femoris muscle strength with a hand-held dynamometer on the affected side in hemiplegic patients. J UOEH. 2004 Mar 1;26(1):1-11. doi: 10.7888/juoeh.26.1. PMID 15038067
- [Background] Taylor NF, Dodd KJ, Graham HK. Test-retest reliability of hand-held dynamometric strength testing in young people with cerebral palsy. Arch Phys Med Rehabil. 2004 Jan;85(1):77-80. doi: 10.1016/s0003-9993(03)00379-4. PMID 14970972
- [Background] Wright RW. Knee injury outcomes measures. J Am Acad Orthop Surg. 2009 Jan;17(1):31-9. doi: 10.5435/00124635-200901000-00005. PMID 19136425

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Structured TENS Therapy | Sham TENS Therapy
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Structured TENS Therapy | Sham TENS Therapy | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (9.0) | 53.3 (7.0) | 50.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Patient's Perception of Pain in the Early Post-operative Period While Utilizing Structured TENS Therapy.
Description: The patient participant will record pain levels during the immediate post-op 2-week time period every day. Day 0 is pain level before surgery. Pain perception measured on a scale from 0-10 with 0 representing no or lowest level pain and 10 representing the highest level of pain
Time Frame: Two weeks postoperatively.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on 0-10 pain level scale
Arm/Group | Structured TENS Therapy | Sham TENS Therapy
Number analyzed (Participants) | 9 | 9
score on 0-10 pain level scale
  Day 0 | 5.10 [3.16 to 7.04] | 5.24 [3.25 to 7.22]
  Day 1 | 4.68 [2.81 to 6.56] | 4.07 [2.19 to 5.95]
  Day 2 | 3.41 [1.54 to 5.28] | 3.28 [1.41 to 5.15]
  Day 3 | 2.78 [0.91 to 4.66] | 2.95 [1.09 to 4.82]
  Day 4 | 2.49 [0.62 to 4.37] | 3.22 [1.36 to 5.09]
  Day 5 | 3.00 [1.13 to 4.88] | 3.26 [1.40 to 5.13]
  Day 6 | 2.20 [0.33 to 4.07] | 2.72 [0.85 to 4.59]
  Day 7 | 2.42 [0.55 to 4.29] | 2.78 [0.92 to 4.65]
  Day 8 | 3.12 [1.25 to 5.00] | 2.63 [0.77 to 4.50]
  Day 9 | 2.59 [0.72 to 4.46] | 2.35 [0.48 to 4.21]
  Day 10 | 2.85 [0.97 to 4.72] | 2.30 [0.44 to 4.17]
  Day 11 | 2.62 [0.75 to 4.49] | 2.93 [1.06 to 4.79]
  Day 12 | 2.50 [0.62 to 4.37] | 2.66 [0.78 to 4.54]
  Day 13 | 2.42 [0.53 to 4.31] | 3.02 [1.13 to 4.91]
  Day 14 | 2.33 [0.41 to 4.25] | 3.20 [1.27 to 5.13]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Transcutaneous Electrical Nerve Stimulation (TENS) therapy is considered an appropriate non-pharmacologic adjunct for the treatment of symptomatic knee arthritis. Since the electrical stimulation applied is minimal, the participants were at no risk of adverse events.
Arm/Group | Structured TENS Therapy | Sham TENS Therapy
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-04-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT01528228/Prot_SAP_000.pdf
  • Informed Consent Form (2011-04-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT01528228/ICF_001.pdf